CLINICAL TRIAL: NCT02889926
Title: Utility of Samples in Bacteriological Prospective Series of Ulcers Leg Infected Clinically
Acronym: ULCERINFECTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ULCERINFECTE
Record Dates: First submitted 2016-08-23; First posted 2016-09-07 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Leg Ulcer
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a swab according to the method of Levine (Experimental)
  Interventions: Biological: a swab according to the method of Levine
- Bacteriological referred to biopsy (Experimental)
  Interventions: Biological: Bacteriological referred to biopsy

INTERVENTIONS:
Biological: a swab according to the method of Levine — A swab according to the method of Levine: choose the pathological area by pressing the swab over the area, with a rotation supported on at least 1 cm² for 5 seconds, to well up from the liquid.
  Arms: a swab according to the method of Levine
Biological: Bacteriological referred to biopsy — Bacteriological referred to biopsy: (This is the hole protocol) Choose the pathological area, debridement of the wound to the pad and a scalpel, cleaning with betadine followed by rinsing with saline, local anesthesia with xylocaine, 6 mm punch for drawing a carrot, put into a sterile container
  Arms: Bacteriological referred to biopsy

SUMMARY:
Leg ulcers are defined as wounds lasting for more than a month. They would receive 0.2% of the population of Western countries. In Europe, the cost per episode of leg ulcers is estimated at 6650 euros (10 000 euros for a foot ulcer). The cost of treatment of wounds would be 2 to 4% of the health budget. Infection is the most common complication of chronic wounds: in most cases, it results in delayed healing, at most, it can result in amputation or serious general complications Bacterial contamination of ulcers is constant. Over time for over 25 years, various studies have shown about relatively identical results. The bacteria are present in over 90% of the etiology of venous leg ulcers. These bacteria are divided into four most common classes: Staphylococcus aureus, Enterococcus, Streptococcus, Pseudomonas. The bacterial ecology changes over time. Indeed Staphylococcus aureus appears first, while the Pseudomonas is associated with ulcers lasting for several months. Anaerobic more difficult to find, are found in 30% of cases Cohabitation between leg ulcers and bacteria often without clinical consequence: These are the stages of infection and colonization.

The infection is related to the proliferation of bacteria and their invasion into the skin, by increasing their virulence (virulence genes acquisition). The increase in the number of bacteria and the multiplicity of bacterial genera are one reason for the increased virulence of bacteria. When bacteria proliferate, because the host defenses are inadequate, or because there is a vascular disease which promotes the proliferation, clinical signs appear

DETAILED DESCRIPTION:
RESEARCH PROJECT Vascular medicine at St Joseph, the management of chronic wounds concerns 80% of hospitalized patients, more than 1,000 patients per year. The reason for hospitalization of these patients outside of revascularization gestures, often performing a skin graft. The existence of an infection of the ulcer on arrival in the service is not a cons-indication for transplant, but will delay it until the signs of infection are brought under control. This scenario is common. The Medical Information department on six months, noted over 100 patients coded "leg ulcers" principal diagnosis and "soft tissue infections" secondary diagnosis.

The importance of this recruitment and the lack of recommendations for the management of these patients justifies the completion of a clinical and microbiological work Until recent months, at the request of Microbiology, bacteriological referred to biopsy was performed first line when suspected of being infected ulcer. After reading the literature, and because of the invasive nature of this gesture, the evaluation of biopsy compared to the swab in a large patient population seems to necessary to the investigators

The proposed work is randomized blinded for microbiological and observational part for the clinical part, on a prospective series of consecutive carriers of infected leg ulcer patients, regardless of the etiology of leg ulcers, excluding dermohypodermitis complicating acute bacterial leg ulcers, with several objectives:

PRIMARY OBJECTIVE Demonstrate the non-inferiority of the swab compared to biopsy in the management of patients hospitalized for infected leg ulcer

two situations

1. If graft Primary endpoint: time in days between the beginning of hospitalization and the day the transplant can be performed. Indeed, the transplants are performed when the doctor determines that the infection is under control
2. If the patient is not grafted:

Primary endpoint: time between the beginning of hospitalization and the end of the ideal hospitalization (when the clinician believes that the patient can get out)

SECONDARY OBJECTIVES and CRITERIA healing rate of patients at 1 month, 3 months and 6 months bacteriological agreement: between the swab and biopsy Comparing the interest of biopsy compared to the swab: percentage of patients for whom the unblinding was necessary and where the biopsy was more informative than the swab (different bacteria require special treatment) .

levies failure rate when the sample is sterile while the ulcer is infected clinically. The collection of demographic, etiological, nutritional profile, and the collection of various local signs can provide indicators of response to the proposed strategy. This type of study has never been done in the population of leg ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over 18 years
* Hospitalized for a leg ulcer whatever the etiology, vascular medicine
* Having clinical criteria and / or biological that suggest infection
* No opposition to participate in the study

Exclusion Criteria:

* Arterial ulcers requiring revascularization (digging ulcers, tendon or bone exposure, necrosis, toe pressure <50 mmHg)
* Ulcers cancer
* Ulcers with acute bacterial cellulitis: large painful acute red leg
* Poor understanding of the French language
* Major hearing impairment
* Severe cognitive or psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of change of treatment response | Hour 24 and hour 72
  Disappearance of at least two signs of infection from the following:
  1. abundant exudate (dry coverage compresses)
  2. local heat
  3. smelly character
  4. 50% decrease of erythema ulcerous perished And reduction in pain of at least two points on the digital scale
Assessement of the infection statue by medical examination | Day-1 and the Day 1 after release
  The physician will answer on the CRF (Clinical Report Form) by: Yes or no

SECONDARY OUTCOMES:
Assessment of change of the ulcer aspect | At Hour 0 and Hour 48
  Photographs taken on arrival to 48 hours before transplantation where graft and out: proofreading blind to validate a posteriori the clinical criteria

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle LAZARETH, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided